CLINICAL TRIAL: NCT06944405
Title: Implementation for Heart Failure Therapies Post-discharge Followed by CardiOSIgnal at HOME
Acronym: COSI-HOME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Precordior Ltd (Industry)
Collaborators: Eshmoun Clinical Research Center (Network); Sahloul Hospital of Sousse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HF202311
Record Dates: First submitted 2025-04-15; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: heart failure; smartphone detection; mechanocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mechanocardiography (Other): Using mechanocardiography for the detection of signs of heart failure.
  Interventions: Device: Mechanocardiography

INTERVENTIONS:
Device: Mechanocardiography — Using mechanocardiography for the detection of signs of heart failure.

SUMMARY:
CardioSignal technology (mechanocardiography) could enable home follow-up after admission for acute heart failure, thus improving guidline-directed medical therapies for heart failure dose escalation while reducing the logistical constraints and stress associated with frequent hospital visits. The intended purpose is to detect signs of HF in adults (aged 18 years or older and < 85 years)

DETAILED DESCRIPTION:
CardioSignal is a smartphone-based innovation using the smartphone's built-in motion sensors (accelerometer and gyroscope) for measuring heart mechanical motion (seismocardiography and gyrocardiography) when placing the phone on the chest for one minute. Innovation also includes cloud-based data analysis for heart motion signals. CardioSignal is a class IIa medical device (software as a medical device) for detecting atrial fibrillation (Afib) and measuring heart rate and soon detecting heart failure. CardioSignal provides accurate and actionable insights of heart health without the need for additional hardware for everyone and everywhere using their smartphone.

Relevant disease areas include atrial fibrillation, heart failure, and related conditions such as stroke and transient ischemic attack (TIA). The innovation supports long-term monitoring and prevention efforts for high-risk populations, including patients with hypertension, diabetes, sleep apnea, cancer, and those with a history of cardiovascular disease as well as patients discharged after a surgical operation.

The primary user groups are patients at home and healthcare providers at point-of-care. CardioSignal empowers patients to self-monitor heart health easily and affordably, enabling proactive care and improved outcomes across diverse populations, including elderly patients, chronic disease sufferers, and those awaiting specialist care or surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted at emergency room for acute heart failure.
* Patients discharged from emergency room after an episode of acute heart failure.
* Either LVEF>40% or ≤40%, either known or assessed during the index hospitalization (however at least 1/3 of patients are required from each category).
* BNP > 200 pg/ml OR NT-ProBNP > 800 pg/ml
* Patients with connected smartphone.

Exclusion Criteria:

* Patients <18 years and >85 years.
* Pregnant women. lactating woman.
* Previous history of allergic asthma at an early age.
* Patients with a history of pulmonary embolism.
* Cardiorespiratory disorders which may be aggravated by the slight compression of the thorax. (patient with a pacemaker).
* Known allergies for: bisoprolol, ramipril, Entresto, spironolactone, empagliflozine, dapagliflozine.
* The participant's inability to adhere to study procedures or give informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
CardioSignal algorithm in guiding | From enrollment to the end of treatment at 90 days
  STRONG-HF study has shown that intensified up-titration of guideline-directed medical therapy in patients with heart failure significantly lowers mortality, the number of re-hospitalizations and healthcare costs. However, the logistics of patients' follow-up makes it difficult to implement it in every day practice in reality (transportation, involvment of relatives, access to echocardiography and lab tests). CardioSignal solution (medical software application installed on a smartphone using phone sensors - mechanocardiography - for the detection of signs of heart failure) could make it easier to implement providing a reliable, simple and cheap solution, which can be used at the point-of-care for heart failure therapy optimization.

CONTACTS AND LOCATIONS:
Locations (2):
- Tunisia (2):
  - Fattouma Bourguiba University Hospital, Emergency department, Monastir, Monastir Governorate
  - Sahloul Hospital, Emergency department, Sousse, Sousse Governorate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tromp J, Sarra C, Nidhal B, Mejdi BM, Zouari F, Hummel Y, Mzoughi K, Kraiem S, Fehri W, Gamra H, Lam CSP, Mebazaa A, Addad F. Nurse-led home-based detection of cardiac dysfunction by ultrasound: results of the CUMIN pilot study. Eur Heart J Digit Health. 2023 Dec 12;5(2):163-169. doi: 10.1093/ehjdh/ztad079. eCollection 2024 Mar. PMID 38505488
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the task force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC) With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2024 Jan;26(1):5-17. doi: 10.1002/ejhf.3024. Epub 2024 Jan 3. PMID 38169072
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631
- [Background] Haddad F, Saraste A, Santalahti KM, Pankaala M, Kaisti M, Kandolin R, Simonen P, Nammas W, Jafarian Dehkordi K, Koivisto T, Knuuti J, Mahaffey KW, Blomster JI. Smartphone-Based Recognition of Heart Failure by Means of Microelectromechanical Sensors. JACC Heart Fail. 2024 Jun;12(6):1030-1040. doi: 10.1016/j.jchf.2024.01.022. Epub 2024 Apr 3. PMID 38573263
- [Background] Bassi NS, Ziaeian B, Yancy CW, Fonarow GC. Association of Optimal Implementation of Sodium-Glucose Cotransporter 2 Inhibitor Therapy With Outcome for Patients With Heart Failure. JAMA Cardiol. 2020 Aug 1;5(8):948-951. doi: 10.1001/jamacardio.2020.0898. PMID 32374344
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2023 Oct 1;44(37):3627-3639. doi: 10.1093/eurheartj/ehad195. No abstract available. PMID 37622666